CLINICAL TRIAL: NCT03793543
Title: Test-Retest Reproducibility of 18F-DCFPyL PET/CT in the Evaluation of Patients With Metastatic Prostate Cancer - an Interscan Variability and Intraobserver Agreement Study
Brief Title: Test-Retest Reproducibility of 18F-DCFPyL PET/CT in the Evaluation of Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J18127; IRB00174393 (Other: JHM IRB)
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: J18127 PSMA PyL 18F-DCFPyL PET/CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL Injection (Experimental): 9±1 mCi (333±37 MBq) IV injection of 18F-DCFPyL
  Interventions: Drug: 18F-DCFPyL Injection

INTERVENTIONS:
Drug: 18F-DCFPyL Injection — A single dose of 9±1 mCi (333±37 MBq) IV injection of 18F-DCFPyL

SUMMARY:
In this study, the investigators intend to validate 18F-DCFPyL test-retest reproducibility in metastatic lesions, in order to investigate whether it serves as a reliable response assessment tool, both to interpret existing studies and to design future longitudinal trials.

DETAILED DESCRIPTION:
The investigators will image patients with widely metastatic castration-sensitive (CSPC) or castration-resistant prostate cancer (CRPC) using 18F-DCFPyL-PET/CT for detection of tumor burden and perform a lesion-based head-to-head comparison with a subsequent near-term (one to seven days) 18F-DCFPyL-PET/CT follow-up scan, to assess test-retest reproducibility of this second-generation PSMA-targeted compound. Second, as it has not been specifically investigated with this compound before, intra-observer agreement as well as inter-scan variability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* History of histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Patients with metastatic castration-sensitive (CSPC) or castration-resistant prostate cancer (CRPC) with evidence of metastatic disease on conventional imaging with CT or bone scan.
* Prior docetaxel-based chemotherapy is permitted
* Documented metastatic prostate cancer progression as assessed by the treating oncologist with either one or both of the following and has not initiated a new therapy after determination of progression: Rising PSA over a minimum 1-week interval and/or radiographic progression in soft tissue and bone metastases (combination of bony and soft tissue metastases)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Administered a radioisotope ≤5 physical half-lives prior to the date of study PET/CT
* Administered IV X-ray contrast medium ≤24 hours prior to the date of study PET/CT
* Administered oral contrast medium ≤120 hours prior to the date of study PET/CT
* Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Change in number of metastatic lesions detected on on 18F-DCFPyL PET/CT from baseline | Change from baseline to up to 4 weeks
  Change in number of metastatic lesions detected on 18F-DCFPyL PET/CT at baseline with a subsequent near-term 18F-DCFPyL PET/CT scan.
Test the intraobserver agreement as assessed by percentage of scans that are read the same on second read | 3 years
  The scans of every patient completing the 2 imaging time points will be reread by the same reader about 4 weeks after the first reading.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rowe, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Werner RA, Lutje S, Habacha B, Bundschuh L, Higuchi T, Buck AK, Kosmala A, Lapa C, Essler M, Lodge MA, Pienta KJ, Eisenberger MA, Markowski MC, Gorin MA, Pomper MG, Rowe SP, Bundschuh RA. Test-retest repeatability of organ uptake on PSMA-targeted 18 F-DCFPyL PET/CT in patients with prostate cancer. Prostate. 2023 Sep;83(12):1186-1192. doi: 10.1002/pros.24577. Epub 2023 May 21. PMID 37211963
- [Derived] Werner RA, Habacha B, Lutje S, Bundschuh L, Higuchi T, Hartrampf P, Serfling SE, Derlin T, Lapa C, Buck AK, Essler M, Pienta KJ, Eisenberger MA, Markowski MC, Shinehouse L, AbdAllah R, Salavati A, Lodge MA, Pomper MG, Gorin MA, Bundschuh RA, Rowe SP. High SUVs Have More Robust Repeatability in Patients with Metastatic Prostate Cancer: Results from a Prospective Test-Retest Cohort Imaged with 18F-DCFPyL. Mol Imaging. 2022 Feb 23;2022:7056983. doi: 10.1155/2022/7056983. eCollection 2022. PMID 35283693